CLINICAL TRIAL: NCT04159571
Title: QuitFast: Evaluating Transcranial Magnetic Stimulation as a Tool to Reduce Smoking Directly Following a Quit Attempt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Virginia Tech Carilion School of Medicine and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00061841
Record Dates: First submitted 2019-11-04; First posted 2019-11-12 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Smoking; Smoking Cessation; Craving; Addiction; Addiction Nicotine; Nicotine Dependence; Cigarette Smoking
Keywords: Transcranial Magnetic Stimulation; Brain Stimulation; Treatment; Neuroimaging
MeSH Terms: conditions — Smoking; Smoking Cessation; Behavior, Addictive; Tobacco Use Disorder; Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Real TBS to the vmPFC (Experimental): Ten sessions of real Theta Burst Stimulation (TBS) will be delivered to the medial prefrontal cortex (mPFC)
  Interventions: Device: Real TBS to the vmPFC
- Sham TBS to the vmPFC (Sham Comparator): Ten sessions of sham Theta Burst Stimulation (TBS) will be delivered to the medial prefrontal cortex (mPFC)
  Interventions: Device: Sham cTBS to the vmPFC

INTERVENTIONS:
Device: Real TBS to the vmPFC — This will be delivered with the Magventure Magpro system; active sham coil (double blinded)
  Arms: Real TBS to the vmPFC
Device: Sham cTBS to the vmPFC — The MagVenture MagPro system has an integrated active sham that uses two surface electrodes placed on the skin beneath the coil.
  Arms: Sham TBS to the vmPFC

SUMMARY:
Cigarette smoking constitutes the greatest preventable cause of mortality and morbidity in the US. The most critical period for long term success of smoking cessation appears to be in the first 7 days after the quit date. A metaanalysis of 3 pharmacotherapy trials revealed that abstinence during the first 7 days was the strongest predictor of 6 month outcomes (n=1649; Odds ratio: 1.4, P <0.0001; Ashare et al. 2013). Prodigious relapse rates during this first week of smoking cessation are likely due to behavioral and neurobiological factors that contribute to high cue-associated craving and low executive control over smoking. The long term goal of the research is to develop evidence-based transcranial magnetic stimulation protocols to facilitate abstinence during this critical period.

DETAILED DESCRIPTION:
The investigators will evaluate the efficacy of TMS to the ventromedial prefrontal cortex (vmPFC) to change smoking-related behaviors. The investigators long-term vision is that TBS would be used as an acute intervention enabling individuals to get through the first week after a smoking quit attempt without relapsing, and transition to more sustainable mechanisms of behavioral change (e.g., medication, cognitive behavioral therapy).

Aim 1 (Strategy 1): Modulating the limbic system as an approach to treatment: vmPFC TBS. Cigarette smokers will be randomized to receive 10 days of real TBS or sham TBS directed to the vmPFC. Intermittently the desire to smoke, and cigarette self-administration will be assessed. The investigators hypothesize that TBS will: 1) decrease the behavioral smoking measures described above, which will be sustained over a time period sufficient to overcome the initial quit attempt (~7-14 days).

The outcomes of the present aims will resolve a critical gap in the investigator's knowledge regarding the efficacy of a promising TMS treatment strategies. These outcomes will be directly translated to a larger longitudinal study evaluating a multi-pronged approach to improving outcomes in traditional pharmacotherapy or behavioral treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (to maximize participation, and minimize effects of cortical atrophy on neuroimaging data)
2. Current cigarette smoker (at least 10 cigarettes per day).
3. Able to read and understand questionnaires and informed consent.
4. Has accommodations within 50 miles of the study site.
5. Is not at elevated risk of seizure (i.e., does not have a history of seizures, is not currently prescribed medications known to lower seizure threshold)
6. Does not have metal objects in the head/neck.
7. Does not have a history of traumatic brain injury, including a head injury that resulted in hospitalization, loss of consciousness for more than 10 minutes, or having ever been informed that they have an epidural, subdural, or subarachnoid hemorrhage.
8. Does not have a history of claustrophobia leading to significant clinical anxiety symptoms.

Exclusion Criteria:

1. Any psychoactive illicit substance use (except marijuana, alcohol, and nicotine) within the last 30 days by self-report and urine drug screen. For marijuana, no use within the last seven days by verbal report and negative (or decreasing) urine THC levels. Participation will be discontinued if participants use psychoactive illicit substances (except nicotine and alcohol) after study initiation.
2. Meets Diagnostic and Statistical Manual of Mental Disorders (DSM)-V criteria for current axis I disorders of major depression, panic disorder, obsessive-compulsive disorder, post traumatic stress syndrome, bipolar affective disorder, schizophrenia, dissociate disorders, eating disorders, and any other psychotic disorder or organic mental disorder.
3. Has current suicidal ideation or homicidal ideation.
4. Has the need for acute treatment with any psychoactive medication including anti-seizure medications and medications for attention-deficit/ hyperactivity disorder.
5. Females of childbearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
6. Has current charges pending for a violent crime (not including DUI related offenses).
7. Does not have a stable living situation.
8. Suffers from chronic migraines.
9. Does not have a stable phone number for contact through calling and/or texting.
10. Does not have a stable means of using WebEx (e.g. personal computer, Internet) for interaction with study personnel during COVID-19.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merideth A. Addicott, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. All data is de-identified.

RESULTS

PARTICIPANT FLOW:
Groups:
- Real TBS to the vmPFC: Ten sessions of real Theta Burst Stimulation (TBS) will be delivered to the left medial prefrontal cortex (mPFC)
  Real TBS to the vmPFC: This will be delivered with the Magventure Magpro system; active sham coil (double blinded)
- Sham TBS to the vmPFC: Ten sessions of sham Theta Burst Stimulation (TBS) will be delivered to the left medial prefrontal cortex (mPFC)
  Sham cTBS to the vmPFC: The MagVenture MagPro system has an integrated active sham that uses two surface electrodes placed on the skin beneath the coil.
Period: Overall Study
Arm/Group | Real TBS to the vmPFC | Sham TBS to the vmPFC
Started | 26 | 14
Completed | 15 | 8
Not Completed | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real TBS to the vmPFC | Sham TBS to the vmPFC | Total
Number analyzed (Participants) | 25 | 13 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (12) | 54 (15) | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 10 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 17 | 11 | 28
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 13 | 38

OUTCOME MEASURES:

1. Primary Outcome: Questionnaire on Smoking Urges Administered Daily Pre TMS to Measure Craving
Description: Questionnaire on Smoking Urges (QSU). This 10-item questionnaire assesses cigarette craving. Participants will be asked to rate from 1 (strongly disagree) to 7 (strongly agree) their agreement with several statements (e.g., "I have a desire for a cigarette right now," and "Nothing would be better than smoking a cigarette right now."). Individual scores can range from 7 to 49. Higher scores represent more craving. QSU scores are averaged per individual per time point. Scores for all time points and all participants were averaged for each arm (real vs sham TMS).
Time Frame: Through study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real TBS to the vmPFC | Sham TBS to the vmPFC
Number analyzed (Participants) | 26 | 14
units on a scale | 16 (8) | 12 (3)

2. Primary Outcome: Self- Report Assessment of Cigarette Use Through Timeline Follow-Back (TLFB) Interview
Description: This self-reported tobacco product use interview asks participants to retrospectively estimate the number of cigarettes they've used each day for the past 30 days or since the previous assessment, whichever is fewer.
Time Frame: Through study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: number of cigarettes per day
Arm/Group | Real TBS to the vmPFC | Sham TBS to the vmPFC
Number analyzed (Participants) | 25 | 13
number of cigarettes per day | 10 (9) | 12 (8)

3. Secondary Outcome: Biochemical Assessment of Tobacco Use Via Quantitative Urine Screens to Detect Cotinine Level
Description: Changes in cigarette use as detected by quantitative cotinine urine screens collected at visits 1, 6, 10, and all follow-ups. Values are averaged across all time points.
Time Frame: Through study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Real TBS to the vmPFC | Sham TBS to the vmPFC
Number analyzed (Participants) | 25 | 13
ng/ml | 1872 (1705) | 1374 (1079)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Real TBS to the vmPFC | Sham TBS to the vmPFC
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/13
Other Adverse Events (participants affected / at risk) | 1/25 | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real TBS to the vmPFC (N=25) | Sham TBS to the vmPFC (N=13)
headache (General disorders) | 1 (1) | 0 (0)
drooping eyelid (General disorders) | 0 (0) | 1 (1)
memory problem (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04159571/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT04159571/ICF_000.pdf